CLINICAL TRIAL: NCT07308457
Title: Comparison of Enhanced Molecular-Level Microbiological Surveillance and Ceftriaxone Prophylaxis in Patients Undergoing Hematopoietic Cell Transplantation: A Randomized, Prospective Medical Experiment
Brief Title: Enhanced Molecular Microbiological Surveillance Versus Ceftriaxone Prophylaxis in Hematopoietic Cell Transplant Patients
Acronym: CRONOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRONOS
Record Dates: First submitted 2025-12-08; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Incidence of Infectious Diseases
Keywords: Hematopoietic Cell Transplantation; Bloodstream Infections
MeSH Terms: conditions — Sepsis | interventions — Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ceftriaxone Prophylaxis (Experimental): Participants assigned to this arm will receive prophylactic ceftriaxone 1 g intravenously once daily, administered at a fixed morning time, starting 24 hours before hematopoietic stem cell infusion (Day -1) and continued until neutrophil recovery or the onset of infection symptoms. All participants undergo continuous body temperature monitoring and standardized microbiological diagnostics in case of fever or suspected infection.
  Interventions: Drug: Ceftriaxone 1000 MG
- No Prophylaxis (No Intervention): Participants in this arm will not receive prophylactic antibacterial therapy. They will undergo the same continuous body temperature monitoring as the intervention group. In case of fever or other indicators of infection, full microbiological diagnostics will be initiated and empirical antibiotic therapy will be started according to clinical judgment and local epidemiology.

INTERVENTIONS:
Drug: Ceftriaxone 1000 MG — Participants in this arm receive prophylactic ceftriaxone administered intravenously at a dose of 1 g once daily. The infusion begins on Day -1 (24 hours before hematopoietic stem cell infusion) and continues until neutrophil recovery (ANC >500/µl for 3 consecutive days) or until signs of infection occur. Ceftriaxone is infused over at least 30 minutes after dissolving 1 g of the drug in 20-40 ml of an intravenous solution that does not contain calcium ions (e.g., 0.9% sodium chloride, 5% glucose, 10% glucose, or other compatible diluents specified in the protocol). Continuous real-time temperature monitoring is performed throughout the intervention period.
  Arms: Ceftriaxone Prophylaxis

SUMMARY:
The goal of this clinical trial is to learn whether close microbiological monitoring without preventive antibiotics works as well as preventive treatment with ceftriaxone in adults receiving stem cell transplants. The study focuses on people with blood cancers or other conditions who need either autologous or allogeneic hematopoietic stem cell transplantation (HSCT).

The main questions the study aims to answer are:

What percentage of participants develop an infection when they do not receive preventive antibiotics compared with those who receive daily ceftriaxone?

Does preventive ceftriaxone lower the chance of specific complications such as bloodstream infections, pneumonia, or severe sepsis?

Researchers will compare two groups:

one group will not receive preventive antibiotics

one group will receive ceftriaxone once a day until their white blood cells recover or until signs of infection appear

All participants will:

have their body temperature monitored continuously starting one day before the transplant

have blood, urine, or other samples collected if they develop fever or symptoms of infection

receive standard medical care during and after the transplant

start standard antibiotic treatment if they develop signs of infection

This study will include 100 adults. The information collected will help determine whether skipping preventive antibiotics is safe in hospitals where bacteria often show resistance to commonly used drugs such as fluoroquinolones.

DETAILED DESCRIPTION:
This study compares two common strategies for preventing infections in adults who receive hematopoietic stem cell transplants (HSCT). People who undergo these transplants often have very low levels of white blood cells for several days or weeks. During this time, they have a high risk of developing serious infections. Many hospitals give preventive antibiotics, but increasing resistance to these drugs has raised questions about whether this approach is still effective.

In this study, participants are randomly assigned to one of two groups. One group receives daily ceftriaxone as preventive treatment. The other group does not receive preventive antibiotics and instead is closely monitored using continuous temperature sensors and frequent microbiological testing. If any participant shows signs of infection, the medical team begins standard antibiotic treatment based on the person's symptoms, test results, and the hospital's local patterns of bacterial resistance.

The study uses modern laboratory methods, including genetic tests to identify bacteria and antibiotic resistance markers. These tests are performed when a participant develops fever or other symptoms of infection. Researchers will track how often infections occur, how severe they are, and whether bacteria are resistant to antibiotics. They will also monitor recovery of blood counts, the length of hospital stay, and whether participants develop complications related to the transplant.

The results of this study may help hospitals choose the safest and most effective approach to preventing infections in transplant patients, especially in settings where resistance to commonly used antibiotics is increasing.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of autologous or allogeneic hematopoietic stem cells from peripheral blood, bone marrow, or cord blood.
* Age ≥18 years.
* Ability to provide written informed consent.
* No active infection for at least 2 weeks prior to transplantation.

Exclusion Criteria:

* Controlled fungal infection.
* Fever of unknown origin.
* Ongoing antibiotic therapy (except cotrimoxazole).
* Participation in any clinical study or experiment at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of infections in the no-prophylaxis group versus the ceftriaxone prophylaxis group | From Day -1 (24h before transplant) until neutrophil recovery (>500/µl for 3 consecutive days)
  The primary outcome is the proportion of patients who develop an infection in the group receiving no antibacterial prophylaxis compared with the group receiving prophylactic ceftriaxone 1 g once daily. Infection is defined in the protocol as the occurrence of: neutropenic fever (single temperature >38.3°C or ≥38.0°C for ≥1 hour with ANC <500/µl or anticipated decline to <500/µl within 48 hours); bloodstream infection/bacteremia confirmed by blood culture; sepsis or septic shock; or clinically/microbiologically confirmed localized infection (respiratory, urinary, gastrointestinal, or other site). Assessment continues until neutrophil recovery (>500/µl for 3 consecutive days).

SECONDARY OUTCOMES:
Incidence of infectious complications | From Day -1 until neutrophil recovery or start of empirical antibiotic therapy (up to ~28 days)
  Proportion of patients experiencing infectious complications defined in the protocol as: neutropenic fever, sepsis, septic shock, pneumonia, sinus infection, urinary tract infection, and gastrointestinal infection. Neutropenic fever is defined as a single temperature >38.3°C or temperature ≥38.0°C for at least one hour with ANC <500/µl or expected decline to <500/µl within 48 hours. Bloodstream infection/bacteremia refers to growth of a microorganism in blood culture with exclusion of contamination. Sepsis and septic shock are defined according to protocol criteria.
Incidence of infections caused by multidrug-resistant pathogens | From Day -1 until neutrophil recovery or start of empirical antibiotic therapy
  Proportion of patients with infections caused by multidrug-resistant pathogens, as determined by microbiological and molecular diagnostics performed at the onset of infection.
Incidence of organ failure | From Day -1 until neutrophil recovery or start of empirical antibiotic therapy
  Proportion of patients who develop organ failure, defined in the protocol as:
  * Respiratory failure: PaO₂ <60 mmHg or PaCO₂ ≥45 mmHg.
  * Circulatory failure: need for vasopressors or inotropes and fluid therapy to maintain systolic blood pressure ≥90 mmHg.
  * Renal failure: acute kidney injury defined as increase in serum creatinine ≥0.3 mg/dl within 48 hours, or ≥1.5-fold increase within 7 days, or urine output <0.5 ml/kg/h for 6 hours.
  * Liver failure: acute hepatic failure <26 weeks with encephalopathy and INR ≥1.5.
Incidence of death | From Day -1 until neutrophil recovery (or earlier if death occurs)
  Proportion of patients who die during the study period in the prophylactic ceftriaxone group compared with the no-prophylaxis group.
Time to neutrophil recovery | From Day -1 until neutrophil recovery
  Time from Day -1 to achievement of neutrophil recovery, defined as three consecutive days with ANC >500/µl.
Time to platelet recovery | From Day -1 until platelet recovery
  Time to achievement of platelet recovery, defined as three consecutive days with platelet count >20,000/µl without platelet transfusions.
Duration of hospitalization | Through hospital discharge (up to approximately 6 weeks)
  Total number of days of hospitalization during the transplant period for each participant.
Incidence and severity of acute graft-versus-host disease (GvHD) | Up to Day 100 after transplantation
  Proportion of patients who develop acute GvHD and its severity, assessed according to MAGIC criteria. Acute GvHD involves skin, liver, and gastrointestinal tract and is evaluated up to Day 100 after transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersytecki zpital Kliniczny nr 1 im. prof. Tadeusza Sokołowskiego Pomorskiego Uniwersytetu Medycznego w Szczecinie, Szczecin, West Pomeranian Voivodeship, Poland